CLINICAL TRIAL: NCT06178471
Title: Safety, Feasibility and Clinical Utility of Critical Care Transesophageal Echocardiography in Hong Kong
Acronym: SAFE-TEE
Status: Not yet recruiting | Type: Observational
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Wincy Wing-Sze Ng, Associate Consultant, Adult Intensive Care Unit, Queen Mary Hospital, Hong Kong
Other Study IDs: 20231212-006-000
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-04

CONDITIONS: Cardiopulmonary Failure
Keywords: Echocardiography; Transesophageal Echocardiography; Critical Care Echocardiography
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — The use of transesophageal echocardiography to diagnose cardiopulmonary failure in ICU patients with suboptimal or inadequate transthoracic echocardiography examinations.

SUMMARY:
Critical care echocardiography is increasingly recognized as an essential skill for intensivists to achieve during their training and fellowship. It serves to provide critical information to guide clinical management in patients with hemodynamic collapse and respiratory insufficiency. While transthoracic echocardiography (TTE) could be adequate for assessment in most situations, patient factors such as body habitus, presence of chest drains and tubes, presence of thoracic surgical dressings, requirement of high ventilatory support may impede operators from obtaining satisfactory images for evaluation. Moreover, operators in TTE require time and experience for adequate skill and technique acquisition. In specific pathologies such as infective endocarditis, presence of thrombus in left atrial appendage, and evaluation of intracardiac shunts, TEE has been shown to be superior to TTE for proper and accurate diagnosis. Therefore, TEE is widely accepted as the preferred and essential modality for echocardiographic examination especially in European countries. Countries such as France and North American have included critical care TEE as a core curriculum in the critical care training pathway.

In Hong Kong, only basic critical care echocardiography using TTE is required during training and in clinical practice. TEE evaluation is mostly performed in cardiac surgery units by cardiac anesthetists and in stable patients by cardiologists. Critical care TEE is seldom performed by intensivists independently for hemodynamic assessment and evaluation of cardiopulmonary failure. This study describes the safety, feasibility, and clinical utility of critical care TEE by critical care fellows in a university-affiliated institute providing tertiary care to the territory. With implementation of this essential technique in a single center, this study serves to act as a generalizable guidance to achieve an ultimate goal of incorporating this technique as core curriculum in critical care training in parts of the world where critical care TEE is not well established.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18; AND
* Admitted to the mixed medical-surgical intensive care units of Queen Mary Hospital in Hong Kong; AND
* Intubated for invasive mechanical ventilation; AND
* Clinically indicated for transesophageal echocardiography (TEE)

Exclusion Criteria:

Patient possessing absolute contraindication(s) to TEE examination according to the ASE guideline 2013:

* Perforated viscus
* Esophageal stricture
* Esophageal tumor
* Esophageal perforation
* Esophageal laceration
* Esophageal diverticulum
* Active upper gastrointestinal bleed

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from cardiopulmonary failure requiring intubation and invasive mechanical ventilation, who benefit from detailed hemodynamic assessment by transesophageal echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Complication of TEE use in the ICU | Within 1 week following the TEE examination
  TEE complications include esophageal perforation, upper gastrointestinal bleeding, loss of artificial airway, oral bleeding, dental injury, odynophagia, mortality

IPD SHARING:
Plan to Share IPD: Undecided